CLINICAL TRIAL: NCT06836219
Title: Measure of Outcomes in Patients With Advanced Ovarian Cancer According to Homologous Recombination Status and Matched Therapies in a Real-world Scenario: A Retrospective and Prospective, Multicenter, Two Cohorts Study
Brief Title: Measure of Outcomes in Patients With Advanced Ovarian Cancer According to Homologous Recombination Status and Matched Therapies in a Real-world Scenario
Acronym: BeLIVE
Status: Recruiting | Type: Observational
Sponsor: Consorzio Oncotech (Other)
Responsible Party: Sponsor
Other Study IDs: BeLIVE
Record Dates: First submitted 2025-01-08; First posted 2025-02-20 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-01

CONDITIONS: Ovarian Cancer
Keywords: Ovarian Cancer; Homologous Recombination status
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort A: Homologous Recombination Deficient (HRD): Homologous Recombination Deficient (HRD) ovarian cancer patients treated with Olaparib plus Bevacizumab as maintenance therapies after partial or complete response to first line platinum-based chemotherapy.
- Cohort B: Homologous Recombination Proficient (HRP): Homologous Recombination Proficient (HRP) ovarian cancer patients treated as for standard clinical practice at clinician's choice.

SUMMARY:
This is a retrospective and prospective, multicenter, observational, two-cohorts study aimed to evaluate clinical outcomes and safety of patients diagnosed with advanced high grade ovarian cancer whose tumor was tested for the homologous recombination (HR) status using a validated HR deficiency test between January 2021 and January 2026.

* Cohort A: Homologous Recombination Deficient (HRD) ovarian cancer patients treated with Olaparib plus Bevacizumab as maintenance therapies after partial or complete response to first line platinum-based chemotherapy.
* Cohort B: Homologous Recombination Proficient (HRP) ovarian cancer patients treated as for standard clinical practice at clinician's choice.

DETAILED DESCRIPTION:
This is a retrospective and prospective, multicenter, observational, two-cohorts study aimed to evaluate clinical outcomes and safety of patients diagnosed with advanced high grade ovarian cancer whose tumor was tested for the homologous recombination status using a validated HRD test between January 2021 and January 2026:

Cohort A: Homologous Recombination Deficient (HRD) ovarian cancer patients treated with Olaparib plus Bevacizumab as maintenance therapies after partial or complete response to first line platinum-based chemotherapy.

Cohort B: Homologous Recombination Proficient (HRP) ovarian cancer patients treated as for standard clinical practice at clinician's choice. Alive patients who have finished the first line treatment (including maintenance) with or without disease progression while signing the informed consent form will be enrolled retrospectively. Alive patients candidate to receive a first line therapy will be enrolledprospectively as soon as molecular data (BRCA status and HRD) are available.

ELIGIBILITY:
Inclusion Criteria:

* Female, age ≥ 18 years at the time of diagnosis
* Patients diagnosed with high-grade serous or endometroid ovarian, fallopian tube, or primary peritoneal cancer undergone to Homologous Recombination test with the MyChoice HRD assay, FoundationOne DX assay or another validated HRD test, between January 2021 and January 2026:

  * Patients with HRD score > 42 or Loss of Heterozygosity (LOH) score high or defined as HR deficient with other tests and treated with Bevacizumab and Olaparib after first line platinumbased chemotherapy will be retrospectively or prospectively enrolled in Cohort A
  * Patients with HRD score < 42 or Loss of Heterozygosity (LOH) score low or defined as HR proficient with other tests and treated with first line platinum-based chemotherapy with or without bevacizumab or others targeted agents will be retrospectively or prospectively enrolled in Cohort B
* Patients must be able to understand the study procedures and agree to participate in the study by providing written informed consent.

Exclusion Criteria:

* Patients who have not performed a validated Homologous Recombination test on tumor sample.
* Patients with germline or somatic BRCA 1 or 2 mutations
* Patients death at the time of inclusion in the current study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Study Population: All patients diagnosed with advanced high grade ovarian cancer who have received a homologous recombination analysis using validated HRD test between January 2021 and January 2026 are eligible. Patients resulted HRD and treated with Olaparib plus Bevacizumab will be included in Cohort A while patient with HRP tumors will be included in the Cohort B. Patients enrolled in the "compassionate use" of Olaparib (CNN program) can be included as well as patients who have received therapies according to clinical practice.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-09-13 (Actual); Primary Completion 2029-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate the clinical outcomes | Until 3 years from enrollment
  The clinical outcomes that will be measured in both study cohorts are:
  progression-free survival (PSF) as the time from treatment's start to disease progression or death for any cause
Evaluate the clinical outcomes | Until 3 years from enrollment
  The clinical outcomes that will be measured in both study cohorts are:
  overall survival (OS) as the time from treatment's start to death for any cause
Evaluate the safety in patients treated with targeted anticancer therapies in each study cohort | Until 3 years from enrollment
  Toxicity evaluated according to CTCAE vers 5.0
Evaluate the safety in patients treated with targeted anticancer therapies in each study cohort | Until 3 years from enrollment
  Percentage of patients with dose reductions
Evaluate the safety in patients treated with targeted anticancer therapies in each study cohort | Until 3 years from enrollment
  Percentage of patients with dose interruptions due to toxicity
Evaluate the safety in patients treated with targeted anticancer therapies in each study cohort | Until 3 years from enrollment
  Percentage of patients with treatment discontinuations due to toxicity
Evaluate the safety in patients treated with targeted anticancer therapies in each study cohort | Until 3 years from enrollment
  Toxicity according to initial dose of targeted agents
Evaluate the safety in patients treated with targeted anticancer therapies in each study cohort | Until 3 years from enrollment
  Incidence of myelodysplastic syndrome and acute myeloid leukaemia in patients receiving PARPi

SECONDARY OUTCOMES:
Describe the clinical outcomes | Until 3 years from enrollment
  according to disease stage
Describe the clinical outcomes | Until 3 years from enrollment
  according to surgical timing
Describe the clinical outcomes | Until 3 years from enrollment
  according to residual disease after surgery in each cohort
Describe the clinical characteristics of patients for which the combination therapy was offered (Cohort A) | Until 3 years from enrollment
  Describe the clinical characteristics of patients for which the combination therapy was offered (Cohort A)
Describe the treatment approach to HRP patients in a real word scenario in Italy (Cohort B) | Until 3 years from enrollment
  Describe the treatment approach to HRP patients in a real word scenario in Italy (Cohort B)

CONTACTS AND LOCATIONS:
Locations (21):
- Italy (21):
  - Istituto Tumori "Giovanni Paolo II" I.R.C.C.S., Bari, BA
  - Azienda Ospedaliero Universitaria di Bologna - Policlinico S.Orsola-Malpighi, Bologna, BO
  - Azienda Ospedaliera S.Croce e Carle Cuneo, Cuneo, CN
  - Azienda Ospedaliera per l'emergenza Cannizzaro, Catania, CT
  - IRCCS Istituto Romagnolo per lo Studio dei Tumori (IRST) "Dino Amadori", Meldola, FC
  - Azienda Ospedaliero Universitario Careggi, Florence, FI
  - IRCCS Policlinico San Martino, Genova, GE
  - Fondazione IRCCS San Gerardo dei Tintori (Monza), Monza, MB
  - Università Vita-Salute San Raffaele (IRCCS San Raffaele - Milano), Milan, MI
  - Istituto Nazionale Tumori (INT) - Milano, Milan, MI
  - Istituto Oncologico Veneto (IOV), Padua, PD
  - Ospedale S. Maria della Misericordia, Perugia, PG
  - Centro di riferimento oncologico - CRO di Aviano, Aviano, PN
  - Istituto Nazionale Tumori Regina Elena - Roma, Roma, RM
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma, RM
  - Ospedale San Paolo - ASL2 - Savona, Savona, SV
  - Ospedale Mauriziano Umberto I, Torino, TO
  - Azienda sanitaria universitaria Friuli Centrale (ASU FC), Udine, UD
  - Azienda Ulss 3 Serenissima, Mestre, VE
  - Istituto Nazionale Tumori IRCCS "Fondazione G. Pascale, Napoli
  - Università degli Studi di Napoli "Federico II", Napoli

DOCUMENTS (1):
  • Study Protocol (2024-02-08): https://cdn.clinicaltrials.gov/large-docs/19/NCT06836219/Prot_000.pdf